CLINICAL TRIAL: NCT03097887
Title: Prospective, Randomized, Controlled Trial of Omega Loop Gastric Bypass With and Without Anti-reflux Sutures - a Pilot Study
Brief Title: Omega Loop Gastric Bypass With And Without Anti-Reflux Sutures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Daniel Moritz Felsenreich, Dr. med. univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1640/2016
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Bile Reflux
Keywords: Omega Loop Gastric Bypass; Reflux; Mini Gastric Bypass
MeSH Terms: conditions — Bile Reflux; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-reflux sutures (Active Comparator): Omega Loop Gastric Bypass with anti-reflux sutures using V-Loc sewing device. Biliary reflux measured using Bilitec 2000™.
  Interventions: Procedure: Omega Loop Gastric Bypass; Device: Bilitec 2000™; Device: V-Loc
- No anti-reflux sutures (Active Comparator): Omega Loop Gastric Bypass without anti-reflux sutures. Biliary reflux measured using Bilitec 2000™.
  Interventions: Procedure: Omega Loop Gastric Bypass; Device: Bilitec 2000™

INTERVENTIONS:
Procedure: Omega Loop Gastric Bypass — Bariatric/metabolic surgical procedure
  Other Names: Mini Gastric Bypass; Single Anastomosis Gastric Bypass
Device: Bilitec 2000™ — The Bilitec 2000™ device will be used to measure the intensity of biliary reflux in the pouch.
Device: V-Loc — Sewing device to perform the anti-reflux sutures.
  Arms: Anti-reflux sutures

SUMMARY:
This proposed trial is designed to answer the following questions: First, is biliary reflux to the distal esophagus present before OLGB and does it increase after the procedure? Second, does performing an OLGB with or without anti-reflux sutures make a difference in (biliary) reflux exposures of the distal esophagus? To answer these questions the investigators plan to perform a randomized, controlled trial involving two groups. Group A will undergo an OLGB without anti-reflux sutures and consists of 50 patients. Group B will receive an OLGB with anti-reflux sutures and also consists of 50 patients.

Gastroscopic evaluation for inflammation and reflux will be performed before and one year after the operation utilizing multilevel intraluminal impedance pH-monitoring (MII-pH) and intragastric Bilitec 2000™. Furthermore, the study will be blinded to the patient. Long-term weight loss, the resolution of comorbidities and the incidence of surgical complications will serve as secondary endpoints. Follow-ups will be performed at 3, 6, and 12 months postoperatively to assess all primary and secondary goals.

DETAILED DESCRIPTION:
Obesity, and especially its comorbidities, has unarguably become the number one threat to human health in the modern world. Western lifestyle leads to an increased prevalence and thus to a higher mortality (i.e. due to cardiovascular diseases).

The positive effects of gastric bypass surgery on excess weight loss and comorbidity resolution are well-known. In contrast to the standard laparoscopic Roux-en-Y Gastric Bypass (RYGB), a newer method, the laparoscopic Omega Loop Gastric Bypass (OLGB), has emerged over the past years. It is believed to be the simpler method involving only one anastomosis (instead of two) and therefore potentially reducing morbidity and mortality whilst maintaining comparable excess weight loss. However, since this new type of gastric bypass is similar to the former Billroth II resection (BII), the carcinoma risk is a concern. The OLGB is different from the BII resection in many ways. For instance, it involves creating an approximately 10 cm long narrow gastric pouch which could prevent the suspected underlying pathogenetic mechanism: biliary reflux to the gastric tube and subsequently to the esophagus. Biliary reflux is suspected to stimulate squamous esophageal cells and Barrett's epithelial cells to produce inflammatory mediators and therefore cause oxidative stress, DNA damage and apoptosis which might lead to adenocarcinoma.

Worldwide, there are currently two different ways to perform an OLGB: with or without anti-reflux sutures, which involve sewing the biliopancreatic limb to the staple line of the pouch using V-Loc (non-absorbable) moving upwards as far as easily possible without creating any tension.

This proposed trial is designed to answer the following questions: First, is biliary reflux to the distal esophagus present before OLGB and does it increase after the procedure? Second, does performing an OLGB with or without anti-reflux sutures make a difference in (biliary) reflux exposures of the distal esophagus?

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 70 years
* Body Mass Index ≥ 35.0 kg/m2
* Exclusion of psychological, endocrinological and anesthesiological contraindications
* Willingness to be assigned to either of the two groups
* Follow-up anticipation
* Willingness to attend all follow-up visits
* Written informed consent

Exclusion Criteria:

* recent or ongoing cardiovascular event within the last 6 months (myocardial infarction, acute coronary syndrome, angioplasty or coronary bypass operation, insult),
* pulmonary embolism or thrombophlebitis within the last 6 months, other bariatric procedures, e.g. gastric banding, Sleeve Gastrectomy, etc., cancer of various origins (exceptions: basal cell carcinoma or carcinoma in situ, disease-free over the last 5 years),
* significant anemia or coagulopathy,
* serum creatinin ≥ 1.5 mg/dl.,
* serum bilirubin or phosphatase elevated or ALT above 3 times the upper limit, stomach, biliopancreatic operations, splenectomy or colon resections, gastric or duodenal ulcer within the last 6 months,
* intraabdominal sepsis (except uncomplicated appendicitis or diverticulitis over 6 months prior to the study),
* organ transplantations,
* anamnestic HIV infection, active TBC, active malaria, chronic Hepatitis B or C, liver cirrhosis,
* alcohol or drug addiction (except caffeine, nicotine) in history,
* acute psychiatric disease interfering with the proposed trial,
* other chronic disease which might interfere with the participation.

Also, patients who are pregnant or plan a pregnancy within the following two years as well as patients who have been included in another study, will be excluded.

Note: Exclusion can be performed by a study coordinator at any time.

Hiatal hernia is not considered an exclusion criterion in this study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Bile Reflux | 1 year
  The primary goal of this study is to assess, whether the choice of method (OLGB with or without anti-reflux sutures) affects the occurrence or severity of biliary reflux to the gastric pouch. Biliary exposure will therefore be assessed before and 12 months after the operation utilizing multilevel intraluminal impedance pH-monitoring (MII-pH) and intragastric Bilitec 2000™.
Bile Reflux | 1 year
  The primary goal of this study is to assess, whether the choice of method (OLGB with or without anti-reflux sutures) affects the occurrence or severity of biliary reflux to the gastric pouch. Extensive biopsies of the gastric pouch and gastroesophageal junction will be taken to prove histological changes due to biliary reflux.

SECONDARY OUTCOMES:
Inflammation | 1 year
  Assessing inflammation before and 12 months after surgery using gastroscopy with biopsy.
Weight loss | 1 year
  Measuring excess weight loss (EWL), to reveal any changes in patients' weight
BMI loss | 1 year
  Excess BMI loss (EBMIL), to reveal any changes in patients' BMI
Complications by point in time/stage | 1 year
  Early postoperative complications (occurring within 30 days) Late postoperative complications (occurring after 30 days)
Complications by severity | 1 year
  Moderate complications (not requiring additional surgical intervention) Severe complications (requiring surgical intervention)
Resolution of hyperlipidemia | 1 year
  Collecting evidence for the resolution of hyperlipidemia
Resolution of hypertension | 1 year
  Collecting evidence for the resolution of hypertension
Resolution of diabetes | 1 year
  Collecting evidence for the resolution of diabetes
Resolution of sleep apnea | 1 year
  Collecting evidence for the resolution of sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prager, Univ. Prof., Study Director — Vienna Medical University
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Analysis will be performed on anonymized data only. A list cross-linking the patient number to the name will be kept secure and is only available to the principal researcher. Written informed consent will be kept for 15 years.